CLINICAL TRIAL: NCT06471660
Title: Influence of Swallowing Impairment on Burden Among Caregivers of Persons With Alzheimer's Disease and Related Dementias
Brief Title: Family Caregiver Online Survey (Dementia and Swallowing Difficulties)
Status: Completed | Type: Observational
Sponsor: University of Oregon (Other)
Collaborators: McMaster University (Other)
Responsible Party: Sponsor
Other Study IDs: STUDY00000738
Record Dates: First submitted 2024-05-24; First posted 2024-06-24 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-06

CONDITIONS: Dementia; Dysphagia; Dementia Alzheimers; Dementia, Vascular; Dementia, Mixed; Dementia With Lewy Bodies; Dementia Frontal; Dementia, Mild; Dementia Moderate; Dementia Severe; Parkinson Disease Dementia; Dementia Frontotemporal
Keywords: caregiver; family caregiver; care partner; survey; remote; virtual; dementia; dysphagia
MeSH Terms: conditions — Dementia; Deglutition Disorders; Alzheimer Disease; Dementia, Vascular; Mixed Dementias; Lewy Body Disease; Lymphoma, Follicular; Pick Disease of the Brain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Family Caregiver Survey is a one-time, 30-minute, online survey for people living with and caring for a family member with dementia. The goal of this research is to explore the needs of family caregivers, specifically when it comes to managing swallowing difficulties (dysphagia).

DETAILED DESCRIPTION:
This research aims to increase our understanding of dysphagia-related caregiver burden and inform the development of a comprehensive dysphagia intervention, one that promotes the health and quality of life of both the caregiver and the person with dementia.

Aim 1. Quantify dysphagia's contribution to burden among family caregivers of persons with dementia across the disease trajectory to identify when may be best to intervene.

Aim 2. Characterize the moderating effects of caregiver readiness and support on dysphagia-related burden and care recipient quality of life to identify what are the most appropriate intervention targets.

ELIGIBILITY:
Inclusion Criteria:

* Be a caregiver for a family member (or chosen family member) with dementia
* Have been caregiving for at least 2 months
* Live at home with the care recipient
* Not be paid for the care provided
* Be over the age of 18
* Live in the US

Exclusion Criteria:

* Not be a caregiver for a family member (or chosen family member) with dementia
* Have been caregiving for less than 2 months
* Not live at home with the care recipient
* Be paid for the care provided
* Be under the age of 18
* Live outside in the US

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Unpaid, adults living with and caring for a family member with dementia with or without swallowing difficulties.
Sampling Method: Non-Probability Sample
Enrollment: 219 (Actual)
Dates: Start 2023-11-07 (Actual); Primary Completion 2025-07-12 (Actual); Study Completion 2025-07-14 (Actual)

PRIMARY OUTCOMES:
Demographic Information | Baseline
  Demographic Questionnaire
Eight-item Informant Interview to Differentiate Aging and Dementia (AD8) | Baseline
  The AD8 is a screening test that is sensitive to detecting early cognitive changes associated with dementia. AD8 is a scale from 0-8, with higher scores signifying more severe cognitive decline.
Global Deterioration Scale (GDS) | Baseline
  The Global Deterioration Scale (GDS) provides an overview of the stages of cognitive function for those suffering from a primary degenerative dementia such as Alzheimer's disease. GDS is a scale from 0-7, with higher scores signifying more severe cognitive decline.
International Dysphagia Diet Standardisation Initiative Functional Diet Scale (IDDSI-FDS) | Baseline
  The IDDSI-FDS is a validated tool that was created in order to capture degree of diet texture restriction. Degree of diet texture restriction has been previously used in the literature as a self- or informant-reported proxy measure for dysphagia severity given that it represents the functional impact of the dysphagia on daily eating. The scale ranges from 0-8, higher scores indicating less diet texture restriction.
Zarit Burden Interview | Baseline
  The Zarit Burden Interview is a valid, reliable, and widely used self-report measure designed to quantify general caregiver burden, incorporating both objective and subjective burden. It queries common areas of concern, including those related to finances, health, social life, and interpersonal relationships, and explores both personal and role strain. Scores range from 0-88, with higher scores signifying more burden.
Caregiver Analysis of Reported Experiences with Swallowing (CARES) | Baseline
  The CARES is a valid and reliable questionnaire designed to screen for dysphagia-related caregiver burden. The 26-item questionnaire explores the potentially burdensome, more objective behavioral and functional changes that have occurred as a result of dysphagia (Part A) and the more subjective stressors experienced by the caregiver (Part B). Scores range from 0-26, with higher scores signifying more dysphagia-related caregiver burden.
Caregiving Competence Scale | Baseline
  The Caregiving Competence Scale, developed for caregivers of persons with dementia and adapted for dysphagia management, is a valid and reliable four-item scale measuring caregivers' perceived adequacy of their own performance. Scores range from 0-12, with higher scores signifying more perceived competence.
Dysphagia-Related Knowledge Questionnaire | Baseline
  The Dysphagia-Related Knowledge Questionnaire is a study-specific measure assessing caregiver knowledge of functional aspects of dysphagia and dysphagia management, including key definitions, signs/symptoms, management techniques, consequences, and the dysphagia trajectory. Scores can range from 0-13, with higher scores signifying more dysphagia-related knowledge.
Preparedness for Caregiving Scale | Baseline
  The Preparedness for Caregiving Scale, adapted for dysphagia management, explores caregivers' perceived preparation related to caring for the physical and emotional needs of their care recipient. Scores range from 0-12, with higher scores signifying more perceived preparedness.
Multidimensional Scale of Perceived Social Support (MSPSS) | Baseline
  The MSPSS is a self-report measure of subjectively assessed social support that has been validated for use within a variety of populations across the lifespan. Scores range from 12-84, with higher scores signifying more perceived social support.
Eating Assessment Tool 10 (EAT-10) | Baseline
  The EAT-10 is a validated, widely used clinically, and easy-to-administer 10-item symptom-specific swallowing outcomes tool designed to understand the extent to which an individual's quality of life has been impacted by dysphagia. While generally completed by patients themselves, previous research has suggested that proxies can reliably report on observable symptoms, such as those rated on the EAT-10 related to swallow function. Scores range from 0-40, with higher scores signifying more severe dysphagia symptoms and greater impact to quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Samantha Shune, Principal Investigator — The University of Oregon
Locations (1):
- Remote study offered by the University of Oregon, Eugene, Oregon, United States